CLINICAL TRIAL: NCT06391164
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of XC243 in Patients With Exacerbation of Chronic Cystitis
Brief Title: Study to Evaluate the Efficacy and Safety of XC243 in Patients With Exacerbation of Chronic Cystitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAIN-XC243-02-01-2023
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cystitis
Keywords: Phase II; VAS
MeSH Terms: conditions — Cystitis

STUDY DESIGN:
Intervention Model Description: Parallel proup
Who Masked: Participant, Investigator
Masking Description: Blinding was carried out by using placebo equivalent to XC243 tablets without active pharmaceutical ingredients (API) and the corresponding labeling of the ID.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- XC243 25 mg (Experimental): XC243 25 mg single
  Interventions: Drug: XC243 25 mg
- XC243 50 mg (Experimental): XC243 50 mg single
  Interventions: Drug: XC243 50 mg
- XC243 75 mg (Experimental): XC243 75 mg single
  Interventions: Drug: XC243 75 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC243 25 mg — Patients will receive the Investigated Product (IP) once in the morning at least 30 minutes before eating for 7-10 days
  Arms: XC243 25 mg
Drug: XC243 50 mg — Patients will receive the IP once in the morning at least 30 minutes before eating for 7-10 days
  Arms: XC243 50 mg
Drug: XC243 75 mg — Patients will receive the IP once in the morning at least 30 minutes before eating for 7-10 days
  Arms: XC243 75 mg
Drug: Placebo — Patients will receive the IP once in the morning at least 30 minutes before eating for 7-10 days
  Arms: Placebo

SUMMARY:
Multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of XC243 in patients with exacerbation of chronic cystitis. It is planned to include patients with chronic cystitis in 4 parallel groups, who will receive XC243 at a dose of 25 mg per day, 50 mg per day, 75 mg per day or placebo for 7-10 days. Efficacy will be assessed by time from first study treatment to resolution of the symptom "Pain, discomfort or burning when urination " assessed on a visual-analog scale (VAS).

DETAILED DESCRIPTION:
The study will be conducted in 8 centers. The study will include the following periods: screening (1 day), treatment period (up to 10 days), follow-up period (7 days).

Upon completion of screening, patients will be randomized to 4 groups in the ratio 1:1:1:1: XC243 at a dose of 25 mg per day, 50 mg per day, 75 mg per day or placebo group.

Also, all patients will be prescribed furasidin daily at the same time, 2 capsules (total dose 100 mg) 3 times a day after meals. On day 8 the investigator will assess the symptoms of cystitis and decide whether to discontinue or prolong a course of therapy with XC243 and furasidin for up to 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of the Form signed and dated by the patient the Patient Information Leaflet informed consent (IMP).
2. Women aged 18 to 65 years inclusive at the time of signing the Informed IMP consent.
3. Established diagnosis of chronic bacterial cystitis (at least three relapses chronic cystitis within 12 months prior to screening or two cases within 6 months prior to screening, including relapse at study entry).
4. The presence of symptoms characteristic of exacerbation of chronic cystitis: pain syndrome (pain in lower abdomen, when urinating), dysuric symptoms (increased urination, pain or burning when urinating, urgency to urinate, feeling of incomplete emptying bladder).
5. The appearance of symptoms of exacerbation of chronic cystitis is not > 48 hours prior to screening visit.
6. Severity of the symptom "Pain, discomfort or burning with urination "from 4 to 8 VAS points.
7. No therapy for current cystitis exacerbation (including phosphomycin and/or furasidin for the treatment of current exacerbation).
8. The patient's consent to refrain from drinking alcoholic beverages during the period of participation in study.
9. Patient consent to use reliable methods contraception throughout the study and through 3 weeks after its end.

Exclusion Criteria:

1. Hypersensitivity to the active and/or any of excipients of the test drug.
2. Hypersensitivity to furasidine and/or any of the excipients concomitant medication.
3. Chronic recurrent cystitis due to infections, sexually transmitted diseases (STIs): gonorrhea, chlamydia, ureaplasmosis, mycoplasmosis, herpes, candidiasis, gardnerellosis, history of trichomoniasis.
4. Chronic recurrent cystitis of viral etiology (caused by adenovirus, cytomegalovirus, virus human papillomavirus herpes).
5. Axillary body temperature ≥ 38 ° C at the screening visit.
6. Presence of menstruation at randomization or estimated onset of menstruation during the period therapy.
7. Pain in the lumbar region.
8. Itching and abundant vaginal discharge and/or purulent discharge from the genitourinary tract.
9. History and/or findings of genitourinary anatomical disorders ultrasound examination (hydronephrosis, sclerosis of the bladder neck, cystocele, descent uterus, paraurethral cyst).
10. Presence of inflammatory diseases of the sexual system (vaginitis, colpitis, cervicitis).
11. Kidney and urinary tract diseases (including urolithiasis), with the exception of chronic cystitis, with a history that, in the opinion of study doctor, may affect the course and results of the clinical study.
12. Chronic renal failure.
13. Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus.
14. History of pseudomembranous colitis.
15. Signs of macrohematuria (admixture of blood in the urine, discoloration of the urine).
16. Previous urinary tract surgery or radiation therapy.
17. History of malignancy, per excluding patients who have not had disease within the last 5 years, patients with completely cured basal cell carcinoma or completely cured carcinoma in situ.
18. Patients with HIV, syphilis, hepatitis B and C diseases, including a history.
19. Liver disease that the study doctor believes may affect course and outcomes clinical trial, history of hepatic failure.
20. Severe, decompensated or unstable somatic diseases (any diseases or conditions that threaten the patient's life or worsen the patient's prognosis, and also make it impossible to conduct clinical trial with this patient).
21. Use of analgesic drugs activity, including systemic NSAIDs, as well as antispasmodic drugs less than 24 hours before taking study drug/placebo.
22. No history of efficacy of furasidine and/or no data furasidin sensitivity based on a history of urine microbiology.
23. The need for the use of drugs from the list of prohibited therapy.
24. Use of systemic antibacterial drugs actions within 7 days prior to screening.
25. Administration of other medicinal products which, in the opinion of the study doctor, may affect progress and results clinical trial.
26. Participation in another clinical trial within 3 months prior to screening.
27. Pregnancy or breastfeeding.
28. Alcohol or drug dependence, history of mental illness.
29. Patient unwillingness or inability to comply with procedures protocol (in the opinion of the study physician).
30. Other conditions that prevent the patient from being included in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time from the first dose of IP treatment until the symptom "Pain, discomfort or burning when urination " disappears (decreases). | Day 1 - Day 10
  Symptom disappears (decreases) criterion "Pain, discomfort or burning during urination "is considered to be the simultaneous fulfillment of the following conditions: Improvement to 1 point or less in VAS and Maintain VAS score of 1 point or less for 24 hours. Within 96 hours (4 days) after the first dose of the IP assessment of the symptom "Pain, discomfort or burning when urinating" will be conducted by the patient after each urination. After 96 hours (from day 5) evaluation this symptom will be carried out 2 times a day (8-00 to 10-00 hours and from 20-00 to 22-00 hours over time).
  Superiority over placebo will be considered established if difference in mean between groups (XC243 - placebo) by symptom reduction time would be greater than 11 hours at the time of treatment evaluation.

SECONDARY OUTCOMES:
Severity of the symptom "Pain, discomfort or burning with urination "as per VAS | Day 1 - Day 11
  Severity of the symptom "Pain, discomfort or burning with urination "as per VAS to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Dynamics of the symptom "Pain, discomfort or burning when urinating" by VAS. | Day 1 - Day 11
  Dynamics of the symptom "Pain, discomfort or burning when urinating" by VAS to End of therapy Visit
Assessment of disease symptoms by Acute Cystitis Symptom Score (ACSS). | Day 1 - Day 11
  ACSS assessment of disease symptoms to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Dynamics of typical symptoms according to the ACSS scale | Day 1 - Day 11
  Dynamics of typical symptoms of the disease according to the ACSS scale to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Dynamics of quality of life according to the ACSS scale | Day 1 - Day 11
  Dynamics of quality of life according to the ACSS scale to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Frequency of patients with disappearance of all typical symptoms diseases | Day 1 - Day 11
  Frequency of patients with disappearance of all typical symptoms diseases (ACSS score 0) to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Time to disappearance of typical disease symptoms for each symptom by ACSS | Day 1 - Day 11
  Time to disappearance of typical disease symptoms (score 0 on the ACSS scale) for each symptom to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Frequency of patients with disappearance of the symptom "pain or urinary burning " by ACSS | Day 1 - Day 11
  Frequency of patients with disappearance of the symptom "pain or urinary burning "(ACSS score 0) to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Frequency of patients with disappearance of the symptom "pain or discomfort in the lower abdomen (suprapubic region) " by ACSS | Day 1 - Day 11
  Frequency of patients with disappearance of the symptom "pain or discomfort in the lower abdomen (suprapubic region) "(score 0 according to ACSS) to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Scale score by Pelvic Pain and Urgency/Frequency Patient Symptom Scale (PUF Scale) | Day 1 - Day 11
  Scale score by PUF Scale to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Dynamics of symptoms of the disease according to the Diary patient. | Day 1 - Day 11
  Dynamics of symptoms of the disease according to the Diary patient to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Dynamics of the symptom "Pain or burning when urinating" according to VAS within first 24 hours post-dose | Day 1 - Day 2
  Dynamics of the symptom "Pain or burning when urinating" according to VAS within first 24 hours post-dose
Mean urinary frequency per day by Patient Diary | Day 1 - Day 11
  Mean urinary frequency per day by Patient Diary to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11)
Assesment by Global Clinical Impression Scale score (CGI-i) | Day 1 - Day 11
  Patient's CGI-i score
Evaluation of the efficacy of therapy by 5 rating scale | Day 1 - Day 11
  Evaluation of the efficacy of therapy by 5 rating scale to Visit 2 (Day 2), Visit 3 (Day 5), Visit 4 (Day 8), End of therapy Visit (Day 11). This scale is assessed by the investigator, where 1 point - absence, 2 points - regression, 3 points - decrease in severity, 4 points - lack of positive dynamics, 5 points - increase in the main clinical symptoms

CONTACTS AND LOCATIONS:
Locations (7):
- Russia (7):
  - Unimed-S Cjsc, Moscow
  - LLC "Research Center Eco-Safety", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic № 112", Saint Petersburg
  - LLC "Clinic Zvezdnaya", Saint Petersburg
  - North-West Center of Evidence-Based Medicine Jsc, Saint Petersburg
  - Prime Rose Medical Center LLC, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 4", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No